CLINICAL TRIAL: NCT06580093
Title: Nutritional Status and Nutritional Problems in Patients With Chronic Kidney Disease Treated With Hemodialysis
Brief Title: Nutritional Status in Patients With Chronic Kidney Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-03363-01; 2022-06295 (Other Grant/Funding Number: The Swedish Research Council)
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Malnutrition
Keywords: Malnutrition; Muscle mass; GLIM
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to investigate how the GLIM criteria* for the diagnosis of malnutrition should be operationalized in patients with chronic kidney disease (CKD) treated with hemodialysis. The main questions it aims to answer are:

* How can malnutrition be defined when applying different combinations and operationalization strategies of the GLIM criteria?
* How can information from other nutrition assessment tools be used in the operationalization of GLIM?
* Which combinations and operationalization strategies of the GLIM criteria can best predict deterioration in quality of life, muscle strength, and increased mortality? An observational study on patients with CKD in hemodialysis will be performed. Variables will be extracted from the Swedish renal registry, SNR and medical records at two hemodialysis units at one university hospital in Sweden. With start in the fall of 2024, data will be collected during two timepoints (baseline and follow-up) when wanted variables for this study are routinely measured at the units.

  * The Global Leadership Initiative on Malnutrition (GLIM) criteria to diagnose malnutrition in adults

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* dialysis duration >3 months prior to recruitment

Exclusion Criteria:

* patients who only have a dialysis frequency of once a week
* patients treated with a combination of peritoneal dialysis and hemodialysis or treated at home
* patients were written consent cannot be obtained due to medical or mental illness or weakened state of health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic Kidney Disease (CKD) treated with hemodialysis at one university hospital in Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Malnutrition diagnosis | From Aug/Sept 2024 to May 2025
  Malnutition diagnosis according to GLIM

SECONDARY OUTCOMES:
Overall survival | From Aug/Sept 2024 to Dec 28
  Overall survival
Muscle strength | From Aug/Sept 2024 to May 2025
  Hand grip muscle strength
Health related quality of life | Aug/Sept 2024 (baseline)
  Health related quality of life according to RAND36
Muscle mass | From Aug/Sept 2024 to May 2025
  Muscle mass according to Bioimpedance Spectroscopy and Calf circumference

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Einarsson, PhD, Principal Investigator — Umeå University
Locations (1):
- Uppsala University hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided